CLINICAL TRIAL: NCT06272331
Title: Postprandial Amino Acid Profiles and Gastric Protein Coagulation After Consumption of Milk and Plant-based Alternatives: an Exploratory Study
Brief Title: Milk and Plant Protein Digestion
Acronym: MAPP-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Principal Investigator, Paul Smeets, Principle Investigator, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NL83162.091.22
Record Dates: First submitted 2024-02-09; First posted 2024-02-22 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Food Digestion
Keywords: Plant-based drink; Milk; Postprandial plasma response; MRI
MeSH Terms: interventions — Milk

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-protein plant-based drink (Other): Ingestion of a low-protein plant-based drink.
  Interventions: Other: Low-protein plant-based drink
- High-protein plant-based drink (Other): Ingestion of a high-protein plant-based drink
  Interventions: Other: High-protein plant-based drink
- Cow's milk (Other): Ingestion of cow's milk.
  Interventions: Other: Cow's milk

INTERVENTIONS:
Other: Low-protein plant-based drink — Ingestion of a low-protein plant-based drink
  Arms: Low-protein plant-based drink
Other: High-protein plant-based drink — Ingestion of a high-protein plant-based drink
  Arms: High-protein plant-based drink
Other: Cow's milk — Ingestion of cow's milk
  Arms: Cow's milk

SUMMARY:
The goal of this study is to explore the effect of protein quantity and quality in plant-based drinks. Healthy normal-weight males aged between 18 and 45 years will be included in the study.

The main objectives are to examine the differences in postprandial amino acid profiles, and to examine differences in gastric behavior between cow's milk and plant based drinks.

Participants will visit after an overnight fast three times and have blood draws before and after consumption one of the study drinks. There will be MRI scans of the stomach before and after consumption of the drink to assess gastric behavior.

DETAILED DESCRIPTION:
Rationale: There is a growing interest in plant-based alternatives for bovine milk. However, these plant-based drinks are not a complete nutritional substitute for bovine milk, especially when focusing on the protein content and quality of these products. Knowledge on the effects of protein quantity and quality of plant based drinks on postprandial plasma responses and gastric behavior compared to bovine milk is lacking.

Objective: To explore the effect of protein quantity and quality of protein in plant-based drinks. In addition, gastric behavior will be examined and compared to that of bovine milk.

Study design: Single-blind randomized cross-over study with three treatments.

Study population: 12 healthy normal-weight males, aged 18-45 y.

Intervention: After an overnight fast, participants will drink cow's milk, or a plant-based drink. Gastric behavior will be monitored using Magnetic Resonance Imaging (MRI). Blood samples will be collected for plasma metabolomic analyses. In addition, wellbeing will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18 - 45 y
* Apparently healthy (self-reported)
* Normal-weight (BMI 18.5 - 25 kg/m2)
* Willing to be informed about incidental findings of pathology
* Willing to comply with the study procedures

Exclusion Criteria:

* Allergy or intolerance for cow milk, lactose or gluten (self-reported)
* Gastric disorders or regular gastric complaints, for example heart burn
* Use of medication which alters the normal functioning of the stomach, such as:

  * Medical drug use that influences the GI tract's normal function, e.g. motility, pH etc.: among others use of protein pump inhibitors, antacids, anti-depressants etc. (judged by study doctor)
  * Medical drug use that influences the GI tract's microbiota: antibiotic use within one month prior to the pre-study screening day (judged by study doctor)
* Following a vegan diet
* Smoking (>2 cigarettes a week)
* Having a chronic illness that could affect food digestion and nutrient absorption including but not limited to kidney disease, thyroid disease and diabetes mellitus (self-reported)
* Alcohol consumption of more than 14 glasses/week
* Having given a blood donation in the past two months
* Hb value below 8.5 mmol/L (as measured with finger-prick method at screening)
* Having a contra-indication to MRI scanning, including, but not limited to:

  * Pacemakers and defibrillators
  * Intraorbital or intraocular metallic fragments
  * Ferromagnetic implants
  * Claustrophobia
* Participating in other research during the study period
* Not having a general practitioner

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Postprandial plasma amino acid profile as characterized by the peak height and iAUC | 5 hours
  Change in postprandial plasma amino acid profile over time

SECONDARY OUTCOMES:
Gastric behavior | 2 hours
  Change in gastric behavior over time as determined from an abdominal MRI scan
Postprandial plasma response | 5 hours
  Change in postprandial plasma response from baseline over time

OTHER OUTCOMES:
Verbal ratings of wellbeing | 5 hours
  Change in wellbeing from baseline over time on a 100-point scale
MRI markers of digestion | 2 hours
  Change in Magnetization Transfer ratio from baseline over time

CONTACTS AND LOCATIONS:
Overall Officials: Paul Smeets, PhD, Principal Investigator — Wageningen University
Locations (1):
- Human Research Unit - Division of Human Nutrition and Health, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: No